CLINICAL TRIAL: NCT07124494
Title: Evaluation of the Effects of Regional Anesthesia Methods Applied in Total Knee Arthroplasty on Joint Range of Motion in the Postoperative Period and Patient Satisfaction
Brief Title: Regional Anesthesia in TKA: Impact on Postoperative Joint Motion and Patient Satisfaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Yasin Tire, MD, Assoc. Prof. Dr. Yasin Tire, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Study Epidural
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Total Knee Arthroplasty; Postoperative Pain; Regional Anesthesia; Knee Range of Motion; Patient Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Spinal-Epidural Anesthesia (Active Comparator): Postoperative analgesia will be provided via epidural catheter with programmed infusion of bupivacaine .
  Interventions: Procedure: Regional anethesia
- Adductor Canal Block (Active Comparator): Ultrasound-guided adductor canal catheter placement and continuous infusion of bupivacaine .
  Interventions: Procedure: Regional anethesia
- Multimodal Intravenous Analgesia (Sham Comparator): Continuous intravenous tramadol infusion with rescue analgesia as required.
  Interventions: Procedure: Regional anethesia

INTERVENTIONS:
Procedure: Regional anethesia — This single-center, prospective, randomized controlled trial aims to compare the effects of three different postoperative analgesia techniques following spinal anesthesia in patients undergoing total knee arthroplasty (TKA). The study will assess the impact of combined spinal-epidural anesthesia, adductor canal block, and multimodal intravenous analgesia on postoperative knee range of motion (ROM). Secondary outcomes include patient satisfaction, opioid consumption, Oxford Knee Score (OKS), activity levels, and visual analog scale (VAS) pain scores.

SUMMARY:
This is a single-center, prospective, randomized controlled trial aiming to evaluate the effects of different regional anesthesia/analgesia techniques on postoperative knee range of motion (ROM) and patient satisfaction following total knee arthroplasty (TKA). Ninety patients undergoing elective TKA under spinal anesthesia will be randomly assigned to one of three groups: 1) spinal anesthesia with epidural catheter, 2) spinal anesthesia followed by adductor canal catheterization, and 3) spinal anesthesia with multimodal intravenous analgesia. The primary outcome is postoperative knee joint ROM measured on postoperative days 1, 2, and 3. Secondary outcomes include patient satisfaction, Oxford Knee Score, postoperative opioid consumption, and VAS scores. The study is conducted at Konya City Hospital and will be completed over a 6-month period.

ELIGIBILITY:
* Minimum Age: 18 Years
* Maximum Age: None
* Sex: All
* Gender Based: No
* Accepts Healthy Volunteers: No
* Inclusion Criteria:

  * Scheduled for primary total knee arthroplasty
  * Age ≥ 18 years
  * American Society of Anesthesiologists (ASA) physical status I-III
  * Accepting neuraxial anesthesia
* Exclusion Criteria:

  * Skin infection at the planned injection site
  * Sepsis
  * Coagulopathy
  * Refusal of neuraxial anesthesia
  * Severe hypovolemia
  * Demyelinating central nervous system disease
  * Age under 18 years
  * Illiterate in Turkish
  * Non-cooperative patients
  * Known allergy or hypersensitivity to bupivacaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Postoperative Knee Range of Motion (ROM) | Postoperative day 1, day 3, day 7, and day 90 after surgery.
  Knee joint flexion and extension range of motion will be measured using a standard goniometer by a blinded assessor. Measurements will be performed with the patient in a supine position, ensuring standardized positioning for all participants.

SECONDARY OUTCOMES:
Total Opioid Consumption | From the end of surgery to 72 hours postoperatively.
  Cumulative opioid consumption (intravenous and oral) will be recorded and converted to morphine milligram equivalents (MME).
Oxford Knee Score (OKS) | Preoperatively (baseline) and postoperative day 90.
  Oxford Knee Score (OKS) questionnaire: Functional outcome will be evaluated using the Oxford Knee Score, a validated 12-item questionnaire assessing pain and physical function.To assess knee pain and functional ability from the patient's perspective.
  Number of questions: 12
  Score range: 0 to 48
  Interpretation:
  0 points = worst possible outcome (severe pain and poor function)
  48 points = best possible outcome (no pain and full function)
  Direction: Higher scores indicate better outcomes
Visual Analog Scale (VAS) Pain Score | Postoperative day 1, day 3, and day 7 after surgery.
  Pain intensity at rest and during movement will be assessed using a 10-cm visual analog scale (0 = no pain, 10 = worst possible pain).
Incidence of Adverse Events Related to Anesthesia or Analgesia | Intraoperative period and up to 90 days postoperatively.
  The occurrence of anesthesia- or analgesia-related complications (e.g., motor weakness, sensory deficits, infection at catheter site, nausea/vomiting, hypotension) will be recorded.
Patient Satisfaction Score | Postoperative day 3 and day 90 after surgery.
  Patient satisfaction with postoperative analgesia will be assessed using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Yasin Tire, Konya, Meram, Turkey (Türkiye)